CLINICAL TRIAL: NCT00382174
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Response Study of the Safety and Efficacy of Thymosin Beta 4 in the Treatment of Patients With Pressure Ulcers
Brief Title: Study of Thymosin Beta 4 in Patients With Pressure Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RegeneRx Biopharmaceuticals, Inc. (Industry)
Responsible Party: David Crockford, VP, Clinical and Regulatory Affairs, RegeneRx Biopharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSPU
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2010-02-01 (Estimated); Last update posted 2010-02-01 (Estimated); Status verified 2010-01

CONDITIONS: Pressure Ulcers
Keywords: pressure ulcers; cutaneous wound- healing; chronic wound-healing; Thymosin Beta 4; laminin-5
MeSH Terms: conditions — Pressure Ulcer | interventions — thymosin beta(4)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): 0.00% thymosin beta 4 w/w administered topically once daily for up to 84 days
  Interventions: Drug: Placebo
- 2 (Active Comparator): 3 doses of thymosin beta 4: 0.01% w/w, 0.02% w/w, and 0.1% w/w, administered topically once daily for up to 84 days
  Interventions: Drug: Thymosin Beta 4

INTERVENTIONS:
Drug: Placebo — Topical administration of 0.00% thymosin beta 4 qd up to 84 days
  Arms: 1
Drug: Thymosin Beta 4 — Topical Administration of 0.01, 0.02, and 0.1% thymosin beta 4 gel qd for up to 84 days
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and effectiveness of Thymosin Beta 4 administered topically in patients with Pressure Ulcers

DETAILED DESCRIPTION:
The purpose of this double-blind, placebo-controlled, dose-escalation study is to evaluate the safety, tolerability and effectiveness of Thymosin Beta 4 (Tβ4), administered topically, in patients with Pressure Ulcers (PU). PU is caused by prolonged pressure or rubbing of the body in areas prone to moisture and friction. PU affects primarily elderly, bedridden patients. Tβ4 is a synthetically-produced copy of a naturally-occurring 43 amino acid peptide that has wound healing and anti-inflammatory properties and can up-regulate the expression of laminin-5.

ELIGIBILITY:
Inclusion criteria:

* Informed Consent Form signed by the patient or patient's legal representative
* Inpatients and outpatients
* At least 1 PU with full-thickness skin loss and no joint capsule or bone exposure
* Surface area between 5 and 70 cm2
* Ulcer present and stable for at least 1 month before enrollment

Exclusion Criteria:

* Use of any experimental drug, or participation in any clinical study, within the 60 days before enrollment
* Use of immunotherapy, or cytotoxic chemotherapy within the 60 days before enrollment. Systemic steroids not allowed 30 days prior to enrollment. Topical therapy other than steroidal is allowed up to 7 days prior to enrollment
* History of adverse events to any ingredients of study medication
* Neurological, cardiovascular, respiratory, hepatic, renal, or metabolic disease likely to interfere with the patient's participation in or completion of the study
* Arterial or venous disorder resulting in ulcerated wounds
* Diabetes mellitus except if disease is determined to be under control with a glycosylated hemoglobin ≤8.5% of total hemoglobin
* Pregnancy or breastfeeding during the study. (A serum pregnancy test will be performed at Screening for female patients of childbearing potential.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry Treadwell, MD, Principal Investigator — Institute for Advanced Wound Care
Locations (12):
- United States (12):
  - Institute for Advanced Wound Care, Montgomery, Alabama
  - Impact Clinical Trials, Beverly Hills, California
  - Long Beach VAMC, Long Beach, California
  - Bay Pines VA Medical Center, Bay Pines, Florida
  - A+ Research, Inc., Miami, Florida
  - Mount Dora Research Center, Inc., Mt. Dora, Florida
  - Hines VAMC, Hines, Illinois
  - Wound Healing Laboratory Plastic Surgery UMass Medical Center, Worcester, Massachusetts
  - New York Presbyterian Hospital, New York, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - New Bridge Medical Center, Warren, Pennsylvania
  - Mcguire VA Medical Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in 2005 and ended in 2008 using 13 sites: Medical Center Clinics, Wound Care Center, Veteran Administration Centers, and Clinical Research Centers.
Pre-assignment Details: Prior to randomization, patients needed to meet specific inclusion and exclusion criteria: results of pregnancy tests needed to be negative; glycosylated hemoglobin tests needed to be less or equal to 8.5% of the total hemoglobin.
Groups:
- Placebo: 0.00% Thymosin Beta 4 (Tβ4), weight/weight (w/w)
- Tβ4 at 3 Doses: 0.01% Tβ4,w/w 0.02% Tβ4,w/w 0.1% Tβ4,w/w
- Placebo vs. Thymosin Beta 4 at 3 Doses: Placebo dose 0.00% thymosin beta 4 vs. thymosin beta 4 at 0.01%, 0.02% and 0.1%
Period: Overall Study
Arm/Group | Placebo | Tβ4 at 3 Doses | Placebo vs. Thymosin Beta 4 at 3 Doses
Started | 18 | 54 | 72
Completed | 14 | 37 | 51
Not Completed | 4 | 17 | 21
Not completed — Lost to Follow-up | 1 | 4 | 5
Not completed — Adverse Event | 1 | 4 | 5
Not completed — Withdrawal by Subject | 1 | 4 | 5
Not completed — Non compliance | 1 | 0 | 1
Not completed — Physician Decision | 0 | 2 | 2
Not completed — Failed to meet criteria | 0 | 1 | 1
Not completed — Wounds merged | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tβ4 at 3 Doses | Total
Number analyzed (Participants) | 18 | 54 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 38 | 55
  >=65 years | 1 | 16 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 14 | 16
  Male | 16 | 40 | 56
Region of Enrollment [Number; unit: participants]
  United States | 18 | 54 | 72

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Thymosin Beta 4 (Tβ4)Applied for up to 84 Days
Description: All Treatment-Emergent Serious Adverse Events (SAEs) and AEs by treatment dose safety population
Time Frame: Up to 84 days
Measure: Number; unit: participants
Arm/Group | Placebo | Tβ4 at 3 Doses | Placebo vs. Thymosin Beta 4 at 3 Doses
Number analyzed (Participants) | 18 | 54 | 72
participants | 18 | 53 | 71

2. Secondary Outcome: Wound Healing Effectiveness of Tβ4 Applied for up to 84 Days
Description: Incidence of wound healing at the end of the study, Day 84
Time Frame: Up to 84 days
Population: Analysis was per protocol,ITT, and using LOCF
Measure: Number; unit: Number of healed participants
Arm/Group | Placebo | Tβ4 at 3 Doses | Placebo vs. Thymosin Beta 4 at 3 Doses
Number analyzed (Participants) | 18 | 54 | 72
Number of healed participants | 3 | 8 | 11

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected for 99 days
Description: AEs were collected at baseline, and weekly thereafter until Day 84 (End of Treatment) and at Day 99.
Arm/Group | Placebo | Tβ4 at 3 Doses | Placebo vs. Thymosin Beta 4 at 3 Doses
Serious Adverse Events (participants affected / at risk) | 5 | 13 | 18
Other Adverse Events (participants affected / at risk) | 13 | 40 | 53
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Tβ4 at 3 Doses | Placebo vs. Thymosin Beta 4 at 3 Doses
Anaemia (Blood and lymphatic system disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Angina (Cardiac disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Chest pain (General disorders) | 1/18 (1) | 1/53 (1) | 2/71 (2)
Pyrexia (General disorders) | 0/18 (0) | 3/53 (3) | 3/71 (3)
Cholecystitis (Hepatobiliary disorders) | 1/18 (1) | 0/53 (0) | 1/71 (1)
Bacteraemia (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Infected Skin Ulcer (Infections and infestations) | 1/18 (1) | 0/53 (0) | 1/71 (1)
Infection (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Lobar pneumonia (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Osteomyelitis (Infections and infestations) | 2/18 (2) | 1/53 (1) | 3/71 (3)
Perianal Abscess (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Pneumonia (Infections and infestations) | 0/18 (0) | 2/53 (2) | 2/71 (2)
Sepsis (Infections and infestations) | 2/18 (2) | 2/53 (2) | 4/71 (4)
Skin infection (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Urinary Tract Infection (Infections and infestations) | 1/18 (1) | 0/53 (0) | 1/71 (1)
Urosepsis (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Wound Infection staphylococcal (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Overdose (Injury, poisoning and procedural complications) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Wound Complications (Injury, poisoning and procedural complications) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Heart Rate Increased (Investigations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Affective Disorder (Psychiatric disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Confusional State (Psychiatric disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1/18 (1) | 0/53 (0) | 1/71 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Tβ4 at 3 Doses | Placebo vs. Thymosin Beta 4 at 3 Doses
Aneamia (Blood and lymphatic system disorders) | 0/18 (0) | 2/53 (2) | 2/71 (2)
Angina Pectoris (Cardiac disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Adreanal Insufficiency (Eye disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Hyperaldosteronism (Endocrine disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Conjunctivitis (Eye disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Dental Caries (Gastrointestinal disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Diarrhea (Gastrointestinal disorders) | 0/18 (0) | 2/53 (2) | 2/71 (2)
Nausea (Gastrointestinal disorders) | 0/18 (0) | 3/53 (3) | 3/71 (3)
Vomiting (Gastrointestinal disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Asthenia (General disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Chest Pain (General disorders) | 1/18 (1) | 1/53 (1) | 1/71 (1)
Chills (General disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Inflammation (General disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Oedema Peripheral (General disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Pyrexia (General disorders) | 1/18 (1) | 8/53 (8) | 9/71 (9)
Cholecystitis (Hepatobiliary disorders) | 1/18 (1) | 0/53 (0) | 1/71 (1)
Hypersensitivity (Immune system disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Abscess (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Bacteraemia (Infections and infestations) | 0/18 (0) | 2/53 (2) | 2/71 (2)
Bacterial Infection (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Beta Haemolytic Streptococcal Infection (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Candidiasis (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Catheter Related Infection (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Catheter Site Infection (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Clostridium Difficile Colitis (Infections and infestations) | 1/18 (1) | 0/53 (0) | 1/71 (1)
Fungal Infection (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Infected Skin Ulcer (Infections and infestations) | 1/18 (1) | 0/53 (0) | 1/71 (1)
Infection (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Lobar Pneumonia (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Nasopharyngitis (Infections and infestations) | 0/18 (0) | 2/53 (2) | 2/71 (2)
Oral Candidiasis (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Osteomyelitis (Infections and infestations) | 2/18 (2) | 2/53 (2) | 4/71 (4)
Otitis Media (Infections and infestations) | 1/18 (1) | 0/53 (0) | 1/71 (1)
Perianal Abscess (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Pneumonia (Infections and infestations) | 0/18 (0) | 3/53 (3) | 3/71 (3)
Sepsis (Infections and infestations) | 2/18 (2) | 5/53 (5) | 7/71 (7)
Skin Infection (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Staphylococcal Infection (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1/18 (1) | 2/53 (2) | 3/71 (3)
Urinary Tract Infection (Infections and infestations) | 4/18 (4) | 9/53 (9) | 13/71 (13)
Urosepsis (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Vaginal Infection (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Wound Infection (Infections and infestations) | 0/18 (0) | 3/53 (3) | 3/71 (3)
Wound Infection Staphylococcal (Infections and infestations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Excoriation (Injury, poisoning and procedural complications) | 0/18 (0) | 2/53 (2) | 2/71 (2)
Joint Injury (Injury, poisoning and procedural complications) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Overdose (Injury, poisoning and procedural complications) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 1/18 (1) | 0/53 (0) | 1/71 (1)
Wound (Injury, poisoning and procedural complications) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Wound Complication (Injury, poisoning and procedural complications) | 1/18 (1) | 4/53 (4) | 5/71 (5)
Wound Secretion (Injury, poisoning and procedural complications) | 0/18 (0) | 2/53 (2) | 2/71 (2)
Blood Albumin Decreased (Investigations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Blood Cholesterol Decreased (Investigations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Blood Potassium Decreased (Investigations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Haematocrit Decreased (Investigations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Haemoglobin Decreased (Investigations) | 1/18 (1) | 1/53 (1) | 2/71 (2)
Heart Rate Increased (Investigations) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Oxygen Saturation Abnormal (Investigations) | 1/18 (1) | 0/53 (0) | 1/71 (1)
Dehydration (Metabolism and nutrition disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0/18 (0) | 2/53 (2) | 2/71 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/18 (0) | 2/53 (2) | 2/71 (2)
Headache (Nervous system disorders) | 0/18 (0) | 2/53 (2) | 2/71 (2)
Muscle Spasticity (Nervous system disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Affective Disorder (Psychiatric disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Anxiety (Psychiatric disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Confusional State (Psychiatric disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Depression (Psychiatric disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Epididymitis (Reproductive system and breast disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1/18 (1) | 0/53 (0) | 1/71 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1/18 (1) | 3/53 (3) | 4/71 (4)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1/18 (1) | 1/53 (1) | 2/71 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Rash (Skin and subcutaneous tissue disorders) | 0/18 (0) | 2/53 (2) | 2/71 (2)
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 1/18 (1) | 0/53 (0) | 1/71 (1)
Skin Maceration (Skin and subcutaneous tissue disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Skin Necrosis (Skin and subcutaneous tissue disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Tooth Extraction (Surgical and medical procedures) | 0/18 (0) | 1/53 (1) | 1/71 (1)
Hypotension (Vascular disorders) | 0/18 (0) | 1/53 (1) | 1/71 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
RegeneRx (RGN) agreements may vary with individual PIs, but will not prohibit any PI from publishing. RGN supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.